CLINICAL TRIAL: NCT01664052
Title: ESS505 Pre-hysterectomy Protocol: Safety and Short Term Effectiveness Study
Brief Title: ESS505 Pre-hysterectomy Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 17035; ESS505-002 (Other: Company internal)
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Contraception

ARMS (2):
- ESS505-A (Essure, BAY1454033) (Experimental): Bilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert with minimal polyethylene terephthalate (PET) fibers (investigational device model ESS505-A) followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement.
  Interventions: Device: ESS505-A (Essure, BAY1454033)
- ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033) (Experimental): Unilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert inclusive of polyethylene terephthalate (PET) fibers (investigational device model ESS505) and contralateral placement of the current commercially approved Essure device, model ESS305 followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement. At the conclusion of the hysterectomy, the uterine cornua and fallopian tubes were sent to a pathology lab for histological preparation, and subsequent evaluation.
  Interventions: Device: ESS505 (Essure, BAY1454033); Device: ESS305 (Essure, BAY1454032)

INTERVENTIONS:
Device: ESS505 (Essure, BAY1454033) — Unilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert inclusive of polyethylene terephthalate (PET) fibers (investigational device model ESS505) followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement. At the conclusion of the hysterectomy, the uterine cornua and fallopian tubes were sent to a pathology lab for histological preparation, and subsequent evaluation.
  Arms: ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033)
Device: ESS305 (Essure, BAY1454032) — Unilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert inclusive of polyethylene terephthalate (PET) fibers (investigational device model ESS505) and contralateral placement of the current commercially approved Essure device, model ESS305 followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement. At the conclusion of the hysterectomy, the uterine cornua and fallopian tubes were sent to a pathology lab for histological preparation, and subsequent evaluation.
  Arms: ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033)
Device: ESS505-A (Essure, BAY1454033) — Bilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert with minimal polyethylene terephthalate (PET) fibers (investigational device model ESS505-A) followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement.
  Arms: ESS505-A (Essure, BAY1454033)

SUMMARY:
This study has been designed to evaluate an investigational model of the Essure System for Permanent Birth Control. The investigational device is designed to offer all the advantages of the currently approved device. In addition, the investigational device offers immediate, permanent contraception without a three-month waiting period or 90-day confirmation test. This study has been designed to evaluate the effectiveness of the investigational device in causing tubal occlusion from insert placement through three months of wearing.

DETAILED DESCRIPTION:
This study has previously been posted by Conceptus, Inc. (US).

After acquiring Conceptus, Inc., Bayer HealthCare AG (Germany) is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are scheduled to undergo a Laparoscopically Assisted Vaginal Hysterectomy (LAVH), Total Abdominal Hysterectomy (TAH), Total Vaginal Hysterectomy (TVH), Total Laparoscopic Hysterectomy (TLH) with Bilateral Total Salpingectomy or Bilateral Salpingo-oophorectomy (BSO), or Laparoscopic Supracervical Hysterectomy (LSH)
* Subjects who are 18 years of age and older
* Subjects who are able and willing to provide written informed consent
* Subjects who agree to use a contraceptive method following Essure placement until the hysterectomy procedure

Exclusion Criteria:

* Subjects with bilateral proximal tubal occlusion
* Subjects who have undergone fallopian tube sterilization
* Subjects with known endometrial or myometrial pathology which is likely to prevent access to the fallopian tube ostia
* Subjects who are post-menopausal
* Subjects with pelvic inflammatory disease (PID)
* Subjects with gynecologic malignancy
* Pregnancy or suspected pregnancy
* Delivery or termination of a pregnancy less than 6 weeks before Essure micro-insert placement
* Known allergy to contrast media
* Any general health condition that may represent, in the opinion of the Investigator, an increased potential risk associated with participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Regina, Saskatchewan, Canada
- Chihuahua City, Chihuahua, Mexico

REFERENCES:
- [Background] Thiel J, Rattray D, Cher DJ. Pre-hysterectomy assessment of immediate tubal occlusion with the third-generation ESSURE insert (ESS505). J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):1055-60. doi: 10.1016/j.jmig.2014.04.020. Epub 2014 May 24. PMID 24861649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 participants were enrolled in two centers.
Period: Phase 1
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033)
Started | 31 (Screening and enrollment) | 0
Insert Placed in at Least One Tube | 25 | 0
HSG 1 Hour Post Placement | 24 | 0
Repeat HSG and Hysterectomy at 30 Days | 9 | 0
Repeat HSG and Hysterectomy at 60 Days | 8 | 0
Repeat HSG and Hysterectomy at 90 Days | 7 | 0
Completed | 24 | 0
Not Completed | 7 | 0
Not completed — No device placement | 6 | 0
Not completed — No HSG 1 hr post placement | 1 | 0
Period: Phase 2
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033)
Started | 0 (Screened and enrolled) | 35
Insert Placed | 0 | 31
HSG 1 Hour Post Placement | 0 | 31
Repeat HSG and Hysterectomy at 30 Days | 0 | 10
Repeat HSG and Hysterectomy at 60 Days | 0 | 10
Repeat HSG and Hysterectomy at 90 Days | 0 | 10
Completed | 0 | 31
Not Completed | 0 | 4
Not completed — No device placement | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- ESS505-A: Bilateral placement of Essure 505A (BAY1454033) insert (with minimal PET fiber).
- ESS305/ESS505: Unilateral placement of Essure 505 (BAY1454033) insert (PET-inclusive) and Contralateral placement of the current commercial Essure device Essure 305 (BAY1454032)
- Total: Total of all reporting groups
Arm/Group | ESS505-A | ESS305/ESS505 | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Mean (Full Range); unit: Years] | 42 [31 to 49] | 40 [28 to 52] | 41 [28 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 66
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Occluded Fallopian Tubes 60 Minutes After Placement of the Insert as Measured by an HSG Evaluation
Description: Hysterosalpingogram (HSG) is an x-ray of the uterus and fallopian tubes after the injection of a contrast material (dye). This test evaluates tubal occlusion.
Time Frame: 60 minutes after insert placement
Measure: Number; unit: Occluded fallopian tubes
Units Other Than Participants: Fallopian tubes
Groups:
- ESS505 (Essure, BAY1454033): Unilateral hysteroscopic placement of the permanent birth control system, Model ESS505 insert inclusive of polyethylene terephthalate (PET) fibers (investigational device model ESS505) and contralateral placement of the current commercially approved Essure device, model ESS305 followed by tubal occlusion evaluation by hysterosalpingogram (HSG) approximately 60 minutes following insert placement. A subsequent HSG was performed prior to the subjects' scheduled hysterectomy procedures at 30 (group 3), 60 (group 2) or 90 days (group 1) post insert placement. At the conclusion of the hysterectomy, the uterine cornua and fallopian tubes were sent to a pathology lab for histological preparation, and subsequent evaluation.
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS305 (Essure, BAY1454032) | ESS505 (Essure, BAY1454033)
Number analyzed (Participants) | 24 | 31 | 31
Number analyzed (Fallopian tubes) | 39 | 31 | 29
Occluded fallopian tubes
  ESS505-A | 36 | NA — ESS505-A not investigated in this group | NA — ESS505-A not investigated in this group
  ESS305 | NA — ESS305 not investigated in this group | 3 | NA — ESS305 not investigated in this group
  ESS505 | NA — ESS505 not investigated in this group | NA — ESS505 not investigated in this group | 28

2. Primary Outcome: Number of Occluded Fallopian Tubes 30 Days Following Placement as Measured by an HSG Evaluation
Description: Hysterosalpingogram (HSG) is an x-ray of the uterus and fallopian tubes after the injection of a contrast material (dye). This test evaluates tubal occlusion. ESS505 and ESS505-A inserts are designed with the addition of an articulated hydrogel plug bonded to the distal portion of the insert with surgical grade adhesive and a nitinol support wire that remains inside the distal inner coil.
Time Frame: 30 days after insert placement
Measure: Number; unit: Occluded fallopian tubes
Units Other Than Participants: Fallopian tubes
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS305 (Essure, BAY1454032) | ESS505 (Essure, BAY1454033)
Number analyzed (Participants) | 9 | 10 | 10
Number analyzed (Fallopian tubes) | 15 | 10 | 10
Occluded fallopian tubes
  ESS505-A | 15 | NA — ESS505-A not investigated in this group | NA — ESS505-A not investigated in this group
  ESS305 | NA — ESS305 not investigated in this group | 10 | NA — ESS305 not investigated in this group
  ESS505 | NA — ESS505 not investigated in this group | NA — ESS505 not investigated in this group | 10

3. Primary Outcome: Number of Occluded Fallopian Tubes 60 Days Following Placement as Measured by an HSG Evaluation
Description: as for outcome 2
Time Frame: 60 days after insert placement
Measure: Number; unit: Occluded fallopian tubes
Units Other Than Participants: Fallopian tubes
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS305 (Essure, BAY1454032) | ESS505 (Essure, BAY1454033)
Number analyzed (Participants) | 8 | 10 | 10
Number analyzed (Fallopian tubes) | 13 | 10 | 9
Occluded fallopian tubes
  ESS505-A | 12 | NA — ESS505-A not investigated in this group | NA — ESS505-A not investigated in this group
  ESS305 | NA — ESS305 not investigated in this group | 10 | NA — ESS305 not investigated in this group
  ESS505 | NA — ESS505 not investigated in this group | NA — ESS505 not investigated in this group | 9

4. Primary Outcome: Number of Occluded Fallopian Tubes 90 Days Following Placement as Measured by an HSG Evaluation
Description: as for outcome 2
Time Frame: 90 days after insert placement
Measure: Number; unit: Occluded fallopian tubes
Units Other Than Participants: Fallopian tubes
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS305 (Essure, BAY1454032) | ESS505 (Essure, BAY1454033)
Number analyzed (Participants) | 7 | 10 | 10
Number analyzed (Fallopian tubes) | 11 | 10 | 10
Occluded fallopian tubes
  ESS505-A | 10 | NA — ESS505-A not investigated in this group | NA — ESS505-A not investigated in this group
  ESS305 | NA — ESS305 not investigated in this group | 10 | NA — ESS305 not investigated in this group
  ESS505 | NA — ESS505 not investigated in this group | NA — ESS505 not investigated in this group | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after signing the informed consent up to 90 days after insert placement.
Description: The reported adverse events cannot be localized to either intervention for women in receipt of ESS305/ESS505, therefore the observed adverse events were reported in a single arm.
Arm/Group | ESS505-A (Essure, BAY1454033) | ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033)
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35
Other Adverse Events (participants affected / at risk) | 2/31 | 5/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESS505-A (Essure, BAY1454033) (N=31) | ESS 305/ESS 505 (Essure, BAY1454032/Essure, BAY1454033) (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Vaginal laceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sensation of pressure (General disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A PI may be requested to delay results communications up to 18 months following study conclusion or until a summary of all study results initiated by Sponsor (first publication) has been published. Following first publication embargo, sponsor may review results communications for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor may request a postponement of results communications not to exceed 180 days.